CLINICAL TRIAL: NCT05135429
Title: Effect of Bathing on Pain, Sleep and Vital Signs of Premature Babies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Principal Investigator, Ayse Sonay Turkmen, Assoc. Prof, Assoc.Prof., Karamanoğlu Mehmetbey University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Newborn
Record Dates: First submitted 2021-10-04; First posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Preterm
MeSH Terms: conditions — Premature Birth | interventions — Baths

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bathing group (Experimental): Newborn bathing will be done by the same nurse for each newborn in the study group. Since the evening hours are thought to be calmer for the baby bath, the hours between 22:00-24:00 will be chosen. Each newborn will be disinfected with only water beforehand and showered in the sinks used to wash the baby in the clinic. Bath time will be limited to two minutes. Newborns will be dried and dressed immediately after bathing. Monitor probes for monitor follow-ups and blood pressure cuffs will be connected to prevent extra touching during measurements.
  Interventions: Other: Bathing
- control group (No Intervention): Newborns in the control group will not receive any intervention. However, body temperature, pulse, respiration, systolic and diastolic blood pressure, saturation, oxygen demand and N-PASS scores will be evaluated and recorded in accordance with the measurement intervals of the newborns in the study group.

INTERVENTIONS:
Other: Bathing — The data of the study were obtained from premature newborns born at 34 weeks and above, who were hospitalized.
  Arms: Bathing group

SUMMARY:
This study was conducted as a randomized controlled experimental study to determine the effect of bathing given to premature babies on pain, sleep and vital signs. The data of the study were obtained from premature newborns born at 34 weeks and above, who were hospitalized in Selcuk University Hospital Neonatal Intensive Care Unit between 1 June and 31 August 2020. The sample size was determined as 64 premature newborns. "Interview and Observation Form, Neonatal Pain/Agitation, Sedation Scale" was used for data collection. The data were evaluated with the SPSS 21.0 package program using percentage, mean, standard deviation, chi-square, t test, Anova and Tukey advanced analysis test.

The research was carried out in the following order. All permissions were obtained for data collection. Individual characteristics were obtained from family members and recorded in the questionnaire. Before the procedure, the pain levels of the newborns were evaluated and recorded. The status of babies in the study or control group was randomly determined according to the hospitalization day (www.randomizer.com).

The newborns in the study group were given a baby bath. The baby's body temperature, pulse, respiration, systolic and diastolic blood pressure, saturation, oxygen demand, and N-PASS scores were evaluated and recorded by two observers before the bath, at the 15th, 30th and 60th minutes after the bath.

No intervention was given to the newborns in the control group. However, body temperature, pulse, respiration, systolic and diastolic blood pressure, saturation, oxygen demand and N-PASS scores were evaluated and recorded in accordance with the measurement intervals of the newborns in the study group.

Cohen's kappa analysis was performed to assess interobserver agreement. Since the inter-observer agreement was found to be excellent (k=0.85), analysis was performed with an observer evaluation.

All newborns were measured at the same time of the day.

DETAILED DESCRIPTION:
The research will be carried out in the second and third level Neonatal Intensive Care Unit of X University Medical Faculty Hospital. 52 nurses and three neonatologists work in the unit. 12 nurses (in-clinical training nurse, nutrition nurse) work during the day and 10 nurses at night. The average number of babies per nurse for care is three. Second and third level patients are hospitalized in the clinic. The total number of beds is 45, with 36 beds at the third level and nine beds at the second level. The average number of babies admitted to the unit and treated is 55/550 monthly/yearly. (Due to the Covid 19 epidemic, the number of hospitalized patients is less than in previous years.)

Outside the unit, there are mother-baby adjustment rooms where the resting needs of mothers are met. There is no restriction on visiting hours for mothers in the clinic, mothers can see and take care of their babies whenever participants want 24/7. Before the Covid 19 epidemic, fathers had visiting hours, but during the epidemic, father visits were abolished.

The sample size was calculated with the G*Power 3.1.5 program with 95% power and 10% difference at 0.05 significance level. The sample size was determined as 64 newborns, 32 children for each group. At the end of the study, Post Hoc power analysis will be performed in order to determine the adequacy of the number of newborns included in the study. When it is determined that 95% power is reached, the data collection process will be terminated.

Randomization of control and study groups; The status of the children to be included in the study in the control or study group will be determined by using "stratification and randomization methods with blocks", taking into account the hospital registration numbers and gender of the newborns. Accordingly, children will be stratified as "girls and boys" for the gender variable. 32 premature newborns will be included in each of the research groups. Since the newborns and their families do not meet each other during the data collection process, the interaction of the newborns in the study and control groups with each other will be prevented.

ELIGIBILITY:
Inclusion Criteria:

* The gestational age of the baby is 34 weeks and above
* Ability to maintain body temperature
* No contraindication for post-surgical bathing
* Not using any analgesic medication
* Body weight of 2000 g and above
* Baby's oxygen need is less than 30%
* No nutritional intolerance
* Parents' willingness to participate in the research

Exclusion Criteria:

* The gestational age of the premature baby is less than 34 weeks.
* Inability to maintain body temperature
* Contraindication of bathing
* Body weight less than 2000 g
* Oxygen requirement greater than 30%
* Presence of nutritional intolerance
* Contraindication of bathing due to clinical course
* Parents' refusal to participate in the study

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-09-04 (Actual)

PRIMARY OUTCOMES:
Pain Score | 60 minutes
  Evaluation of the change in the pain status of the newborn according to the initial value with Neonatal Pain Agitation And Sedation Scale (N-PASS) just before the bath, 15, 30 and 60 minutes after the bath.
  N-PASS, which consists of two separate sections measuring the sedation level and pain level of the baby; It consists of 5 sub-parameters including crying and restlessness, behavior-state, facial expression, hands and feet, body tension and vital signs. A score between 0 and +2 is given for each behavioral and physiological criterion in the evaluation of pain, and between 0 and -2 in the evaluation of sedation. If the baby was born before 30 weeks of gestation, +1 point is added to the total score in the pain assessment. The total pain score ranges from 0 to +11, and the total sedation score ranges from 0 to 10. A high score indicates that the severity of pain is high.
sleep time | two hours
  Measuring the sleep time of the newborn with a stopwatch evaluation
body temperature | 60 minutes
  Evaluation of the change in the temperature of the newborn according to the initial value with a thermometer 15, 30 and 60 minutes after bathing, just before bathing.
pulse rate | 60 minutes
  Evaluation of the newborn's heart rate 15, 30 and 60 minutes after bathing, with a thermometer just before bathing, according to the baseline value.
respiratory rate | 60 minutes
  Evaluation of the change in the respiratory rate of the newborn at 15, 30 and 60 minutes after the bath, by observation (during 1 minute) just before the bath, relative to the baseline value.
Blood pressure | 60 minutes
  Evaluation of the change in blood pressure of the newborn at 15, 30 and 60 minutes after the bath, with a sphygmomanometer just before the bath, according to the baseline value.
oxygen saturation | 60 minutes
  Evaluation of the change in oxygen saturation of the newborn 15, 30 and 60 minutes after the bath, with a saturation device just before the bath, according to the initial value.

CONTACTS AND LOCATIONS:
Locations (1):
- KaramanogluMehmetbeyU, Karaman, Turkey (Türkiye)